CLINICAL TRIAL: NCT06945224
Title: Trastuzumab-deruxtecan In Metastatic Breast Cancer Patients: A ReaL World Study of Chinese Population
Brief Title: A ReaL World Study of DS-8201
Acronym: EXPLORE
Status: Active, not recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Professor, Fudan University
Other Study IDs: EXPLORE
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Metastatic; Treatment Efficacy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients received DS-8201: HER2-positive and HER2-low breast cancer patients who received DS-8201 in the advanced stage

SUMMARY:
A ReaL world study of DS-8201

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 or above;
2. The Eastern Cooperative Oncology Group (ECOG) physical condition score of the United States is ≤2;
3. HER2 positive (IHC 3+ or IHC 2+ and ISH+) confirmed by tumor histology or cytology, and having received one or more anti-HER2 drug treatments previously; Or low expression of HER2 confirmed by tumor histology or cytology (IHC 1+ or IHC 2+ and ISH-), and having received at least one systemic treatment in the metastatic disease stage previously, or unresectable or metastatic breast cancer that relapsed during adjuvant chemotherapy or within 6 months after the completion of adjuvant chemotherapy;
4. Receive goldtrastuzumab treatment in the advanced stage;
5. During the study period, voluntarily abide by this trial protocol and receive regular follow-ups;
6. All women of childbearing age, fertile men or their spouses who have no plans for fertility or sperm donation throughout the trial period until 6 months after the last dose, or who voluntarily take effective contraceptive measures.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Those with acute or chronic infections, or those with other serious diseases at the same time, are judged by the researchers as unsuitable for this study;
3. Having suffered from other malignant tumors within 5 years (excluding the following situations: cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and papillary thyroid carcinoma; A second primary cancer that has been completely cured and has no recurrence within five years; Researchers have clearly identified which primary tumor source the metastatic foci belong to.
4. Those with mental illness or mental disorders, poor compliance and inability to cooperate and describe treatment responses;
5. Those with severe organic diseases or major organ failure, such as decompensated heart, lung, liver or kidney failure, which makes them unable to tolerate treatment;
6. Patients allergic to trastuzumab;
7. Patients who changed their treatment regimens after trastuzumab treatment due to reasons other than disease progression or intolerable adverse reactions;
8. The researcher believes that the patient has other circumstances that make them unsuitable for participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients who received DS-8201 in the advanced stage
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | Six months after the last patient was enrolled
  PFS was defined as the time interval from the date of DS-8201 initiation until date of progressive disease (PD) or death from any causes, whichever occurred first.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer center, Shanghai, China, China